CLINICAL TRIAL: NCT05205759
Title: Adaptive, Randomized, Non-inferiority Trial to Evaluate the Efficacy of Monoclonal Antibodies in Outpatients With Mild or Moderate COVID-19
Brief Title: Non-inferiority Trial on Monoclonal Antibodies in COVID-19
Acronym: MANTICO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stop for futility after the onset of the omicron wave
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government); Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Evelina Tacconelli, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MANTICO; 2021-002612-31 (EudraCT Number)
Record Dates: First submitted 2022-01-15; First posted 2022-01-25 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Coronavirus Infections; Monoclonal antibodies; Bamlanivimab Etesevimab; Casirivimab Imdevimab; Sotrovimab
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — bamlanivimab and etesevimab drug combination; sotrovimab; casirivimab and imdevimab drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bamlanivimab Etesevimab (Experimental): Bamlanivimab 700 mg + Etesevimab 1400 mg administered in 250 mL prefilled 0.9% sodium chloride injection infusion solution over one hour
  Interventions: Drug: Bamlanivimab Etesevimab
- Sotrovimab (Experimental): Sotrovimab 500 mg administered in 100 mL prefilled 0.9% sodium chloride injection infusion solution over 1/2 hour
  Interventions: Drug: Sotrovimab
- Casirivimab Imdevimab (Active Comparator): Casirivimab 600 mg + Imdevimab 600 mg administered in 250 mL prefilled 0.9% sodium chloride injection infusion solution over one hour
  Interventions: Drug: Casirivimab-Imdevimab

INTERVENTIONS:
Drug: Bamlanivimab Etesevimab — Single intravenous infusion of bamlanivimab 700 mg and etesevimab 1400 mg, administered together [1 bamlanivimab vial (700 mg/20 mL) and 2 etesevimab vials (700 mg/20 mL)] in a 250-mL prefilled 0.9% Sodium Chloride infusion bag over one hour.
  Arms: Bamlanivimab Etesevimab
Drug: Sotrovimab — Single intravenous infusion of sotrovimab 500 mg (500 mg/8 mL), administered in 100 mL prefilled 0.9% sodium chloride injection infusion solution over 1/2 hour.
  Arms: Sotrovimab
Drug: Casirivimab-Imdevimab — Single intravenous infusion of casirivimab 600 mg + imdevimab 600 mg, administered together in 250 mL prefilled 0.9% sodium chloride injection infusion solution over one hour. Casirivimab and imdevimab are each supplied in individual single use vials. Casirivimab is available as 300 mg/2.5 mL (120 mg/mL) or 1332 mg/11.1 mL (120 mg/mL). Imdevimab is available as 300 mg/2.5 mL (120 mg/mL) or 1332 mg/11.1 mL (120 mg/mL).
  Arms: Casirivimab Imdevimab

SUMMARY:
Currently, 3 anti-SARS-CoV-2 monoclonal antibody products have received Emergency Use Authorizations from the Italian Medicines Agency (AIFA) for the treatment of mild to moderate COVID-19 in non hospitalized patients with laboratory-confirmed SARS-CoV-2 infection who are at high risk for progressing to severe disease and/or hospitalization (bamlanivimab plus etesevimab, sotrovimab, and casirivimab plus imdevimab). Differently from casirivimab/imdevimab and sotrovimab, the European Medicines Agency (EMA) has never recommended authorising the combination bamlanivimab/etesevimab for treating COVID-19. Moreover, the evidence on sotrovimab relies on the interim analysis results of an ongoing randomised placebo-controlled clinical trial [1], unlike the combinations bamlanivimab/etesevimab and casirivimab/imdevimab, whose results of the randomised placebo-controlled trials were published after having completed the enrolment [2,3]. The study aims at assessing the non-inferiority of bamlanivimab plus etesevimab and sotrovimab vs. casirivimab plus imdevimab on COVID-19 progression in patients aged at least 50 years at an early stage of the disease. The progression of COVID-19 disease (hospitalization, need for supplementary oxygen therapy at home, death) within 14 days of randomisation is the composite outcome variable on which the calculation of the sample size is based. Based on available data regarding the reduction in the number of hospitalisations and medical visits with the use of casirivimab plus imdevimab at an early-stage of COVID-19, a disease progression of 5% has been estimated in the reference arm. 5% delta margin was considered clinically relevant, taking into account both the estimates of disease progression in the study population in absence of early treatment with monoclonal antibodies (20%, based on national data) and the efficacy of the reference standard. Therefore, 1260 participants will be randomly assigned in an equal ratio between the reference standard and each of the other two experimental arms (1:1:1). Randomization will be computer-generated in permuted blocks with a stratification based on site.

DETAILED DESCRIPTION:
Sample size. The parameters for the sample size estimation were derived from the only double-blind, randomised, placebo-controlled trial assessing the clinical efficacy of casirivimab/imdevimab (reference standard) [3]. Hospitalisation related to COVID-19 or all-cause mortality in this study occurred in 7 of 736 patients in the casirivimab/imdevimab 1200-mg group (1.0%) and in 24 of 748 patients in the placebo group who underwent randomisation concurrently (3.2%) (relative risk reduction, 70.4%; P=0.002). Assuming a non-inferiority margin of 5%, 420 patients per group were needed to achieve 90% power with a 1-sided α level of .025, allowing for 5% dropout. A 5% non-inferiority margin was chosen as the maximal difference between treatments in COVID-19 progression that would be clinically acceptable by consultation with Infectious Diseases and clinical trial specialists involved in the protocol development.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Informed consent by the subject or legally authorized representative
* Laboratory-confirmed SARS-CoV-2 infection, as determined by antigen or nucleic acid identification in any specimen, within 4 days of eligibility assessment
* Peripheral oxygen saturation ≥ 94% on room air and not requiring supplemental oxygen
* Onset of symptoms within 4 days of eligibility assessment. Onset time of symptoms is defined as the time when the patient experienced the presence of at least one of the following SARS-CoV-2 infection-associated symptoms for the first time [4]: cough, nasal congestion, sore throat, feeling hot or feverish, myalgia, fatigue, headache, anosmia/ageusia, nausea, vomiting, and/or diarrhoea

Exclusion Criteria:

* Previously or currently hospitalized or requiring hospitalization
* Respiratory distress with respiratory rate ≥ 25 breaths/min
* Heart rate ≥ 125 beats per minute
* Peripheral oxygen saturation ≤ 93% on room air at sea level
* Known allergies to any of the components used in the formulation of the trial drugs
* Hemodynamic instability requiring use of pressors within 24 hours of randomization
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that could potentially lead to hospitalization within 30 days
* Any co-morbidity requiring surgery within 7 days or that is considered life-threatening within 90 days
* History of positive SARS-CoV-2 test prior to 4 days of the eligibility assessment
* Previous treatment with a SARS-CoV-2 specific monoclonal antibody
* History of convalescent COVID-19 plasma treatment
* Participation in a clinical study involving an investigational intervention within the last 30 days
* Pregnancy or breast feeding
* Investigator site personnel directly affiliated with this study
* Sexually active women of childbearing potential or sexually active men who are unwilling to practice effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose
* Inability to participate to the study follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
COVID-19 progression | 14 days
  (1) hospitalization or (2) need of supplemental oxygen therapy at home or (3) death within 14 days of randomisation

SECONDARY OUTCOMES:
Visits to the Emergency Room | 28 days
  Number of visits to the Emergency Room without subsequent hospitalization within 28 days of randomization
Duration of supplemental oxygen therapy | 90 days
  Days of supplemental oxygen therapy within 90 days of randomization
Duration of hospitalization | 90 days
  Days of any hospitalization within 90 days of randomization
Non-invasive ventilation | 28 days
  Rate of patients undergoing non-invasive ventilation within 28 days of randomization
Duration of non-invasive ventilation | 90 days
  Days of non-invasive ventilation within 90 days of randomization
Mechanical ventilation | 28 days
  Rate of patients undergoing mechanical ventilation within 28 of randomization
Duration of mechanical ventilation | 90 days
  Days of mechanical ventilation within 90 days of randomization
28-day mortality | 28 days
  Death rate at 28 days of randomization
Duration of symptoms | 90 days
  Days of symptoms within 90 days of randomization

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - IRCCS Policlinico di S. Orsola, Bologna
  - PO SS Trinità di Cagliari, Cagliari
  - Azienda Ospedaliera Cannizzaro, Catania
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele, Catania
  - PO Garibaldi Nesima, Catania
  - Azienda Socio-Sanitaria Territoriale di Cremona, Cremona
  - Ospedale S. Maria Annunziata, Florence
  - Covid Hospital Jesolo, Jesolo
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera dei Colli, presidio ospedaliero Cotugno, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - AOU Policlinico, Palermo
  - Azienda Ospedaliera S. Maria della Misericordia, Perugia
  - Università degli Studi di Pescara, Pescara
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Ospedale San Paolo ASL 2 Savonese, Savona
  - AOU Città della Salute e Scienza, Presidio Molinette, Torino
  - Azienda Sanitaria Universitaria Giuliano-Isontina (ASUGI), Trieste
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
  - Azienda Ospedaliera di Verona, Verona

REFERENCES:
- [Background] Gupta A, Gonzalez-Rojas Y, Juarez E, Crespo Casal M, Moya J, Falci DR, Sarkis E, Solis J, Zheng H, Scott N, Cathcart AL, Hebner CM, Sager J, Mogalian E, Tipple C, Peppercorn A, Alexander E, Pang PS, Free A, Brinson C, Aldinger M, Shapiro AE; COMET-ICE Investigators. Early Treatment for Covid-19 with SARS-CoV-2 Neutralizing Antibody Sotrovimab. N Engl J Med. 2021 Nov 18;385(21):1941-1950. doi: 10.1056/NEJMoa2107934. Epub 2021 Oct 27. PMID 34706189
- [Background] Dougan M, Nirula A, Azizad M, Mocherla B, Gottlieb RL, Chen P, Hebert C, Perry R, Boscia J, Heller B, Morris J, Crystal C, Igbinadolor A, Huhn G, Cardona J, Shawa I, Kumar P, Adams AC, Van Naarden J, Custer KL, Durante M, Oakley G, Schade AE, Holzer TR, Ebert PJ, Higgs RE, Kallewaard NL, Sabo J, Patel DR, Dabora MC, Klekotka P, Shen L, Skovronsky DM; BLAZE-1 Investigators. Bamlanivimab plus Etesevimab in Mild or Moderate Covid-19. N Engl J Med. 2021 Oct 7;385(15):1382-1392. doi: 10.1056/NEJMoa2102685. Epub 2021 Jul 14. PMID 34260849
- [Background] Weinreich DM, Sivapalasingam S, Norton T, Ali S, Gao H, Bhore R, Xiao J, Hooper AT, Hamilton JD, Musser BJ, Rofail D, Hussein M, Im J, Atmodjo DY, Perry C, Pan C, Mahmood A, Hosain R, Davis JD, Turner KC, Baum A, Kyratsous CA, Kim Y, Cook A, Kampman W, Roque-Guerrero L, Acloque G, Aazami H, Cannon K, Simon-Campos JA, Bocchini JA, Kowal B, DiCioccio AT, Soo Y, Geba GP, Stahl N, Lipsich L, Braunstein N, Herman G, Yancopoulos GD; Trial Investigators. REGEN-COV Antibody Combination and Outcomes in Outpatients with Covid-19. N Engl J Med. 2021 Dec 2;385(23):e81. doi: 10.1056/NEJMoa2108163. Epub 2021 Sep 29. PMID 34587383
- [Background] U.S. Department of Health and Human Services Food and Drug Administration. Assessing COVID19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment. Available at https://www.fda.gov/regulatory-information/search-fda-guidance-documents/assessing-covid-19-related-symptoms-outpatient-adult-and-adolescent-subjects-clinical-trials-drugs. Accessed 30 March 2022.
- [Derived] Mazzaferri F, Mirandola M, Savoldi A, De Nardo P, Morra M, Tebon M, Armellini M, De Luca G, Calandrino L, Sasset L, D'Elia D, Sozio E, Danese E, Gibellini D, Monne I, Scroccaro G, Magrini N, Cattelan A, Tascini C; MANTICO Working Group; Tacconelli E. Exploratory data on the clinical efficacy of monoclonal antibodies against SARS-CoV-2 Omicron variant of concern. Elife. 2022 Nov 22;11:e79639. doi: 10.7554/eLife.79639. PMID 36413383